CLINICAL TRIAL: NCT03684096
Title: The Effect of the Non-estrogenic Pollen Extract PCC-100 on Hot Flushes During Adjuvant Hormonal Treatment for Breast Cancer in Postmenopausal Women and in Menopausal Women Without a History of Breast Cancer
Brief Title: Effect of Non-estrogenic Pollen Extract PCC-100 on Hot Flushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC/2017/1261
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Hot Flashes; Postmenopausal Symptoms
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-estrogenic pollen extract PCC-100 (Active Comparator): After randomisation patients will be devided in the group who will take the non-estrogenic pollen extract PCC-100 or the group who will receive placebo. The patients will take the drug or placebo for 12 weeks. During these 12 weeks the patients need to register the number and severity of the hot flashes. The patient will have 2 study visits during those 12 weeks.
  Interventions: Dietary Supplement: non-estrogenic pollen extract PCC-100
- placebo (Placebo Comparator): After randomisation patients will be devided in the group who will take the non-estrogenic pollen extract PCC-100 or the group who will receive placebo. The patients will take the drug or placebo for 12 weeks. During these 12 weeks the patients need to register the number and severity of the hot flashes. The patient will have 2 study visits during those 12 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: non-estrogenic pollen extract PCC-100 — non-estrogenic pollen extract PCC-100
  Arms: non-estrogenic pollen extract PCC-100
Other: placebo — placebo -non-estrogenic pollen extract PCC-100
  Arms: placebo

SUMMARY:
Many postmenopausal women have vasomotor symptoms during adjuvant hormonal treatment for breast cancer. PCC-100 is a pollen extract used for alleviation of postmenopausal symptoms. In a randomised, double blinded study pollen extract PCC-100 will be used to treat vasomotor complaints in postmenopausal women under adjuvant hormonal treatment and also in menopausal women without a history of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, between 50 and 65 years old (extremes included) at the time of signing the informed consent form;
* spontaneous amenorrhea for at least 6 consecutive months in combination with a hormonal diagnosis of being postmenopausal (FSH > 40 mU/ml and E2 < 20 pg/ml. In subjects using Tamoxifen, only E2 needs to be determined) or spontaneous amenorrhea for at least 12 consecutive months or having had a bilateral oophorectomy at least 6 weeks prior to screening (with or without hysterectomy);
* a history of breast cancer, whatever the received treatment, and currently taking aromatase inhibitors or Tamoxifen since at least 4 weeks. This criterion is not applicable to the 100 subjects entering the study without a history of breast cancer;
* a minimum of 49 moderate to severe hot flushes or night sweats during 7 consecutive 24-h periods;
* a body mass index [BMI] between 18.0 and 35.0 kg/m2, inclusive;
* proven normal glycaemia and normal thyroid function as evidenced in a recent serum analysis (in the last year) performed by the General Practitioner or gynaecologist;
* The subject is able to understand and comply with the protocol requirements, instructions, and protocol-stated restrictions.

Exclusion Criteria:

* Recently, an abnormal cervical Pap smear that requires surgery within 6 months;
* acute or chronic thromboembolic disease, liver disease and/or renal impairment;
* uncontrolled diabetes mellitus;
* uncontrolled hypertension;
* uncontrolled thyroid disorders;
* the subject has a history of a major depression or post-traumatic stress disorder [PTSD] within 2 years of screening. Women taking antidepressants can be included after a wash out period of 6 weeks;
* use of (non-)hormonal treatments to reduce hot flushes, unless a wash-out period is respected;
* a history or presence of allergy or intolerance to the investigational product or any component of the investigational product or drugs in this class. Or history of drug or other allergy that, in the opinion of the investigator contraindicates subject participation;
* a history of alcohol or substance abuse or dependence in the 12 months before screening as determined by the investigator;
* judged by the investigator to be unsuitable for any reason.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — only women will be recruited
Enrollment: 69 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Daily frequency of hot flashes | 12 weeks
  Daily frequency of hot flashes as mentioned in the daily diary the subjects need to complete during 12 weeks. The patient indicate in the diary the number, intensity (mild, moderate, severe) of hotflashes every day

SECONDARY OUTCOMES:
Menopause symptoms | 6-8 weeks after randomisation and 12 weeks after randomisation
  Symptoms related to menopause will be asked to the patients by using the Menopause Rating Scale (MRS), this is a questionnaire with 11 questions about menopause and you can scale every question from 1 (no complaints) to 4 (severe).
Menopause symptoms | 6-8 weeks after randomisation and 12 weeks after randomisation
  Symptoms related to menopause will be asked to the patients by using the Green Climacteric Scale. This is a questionnaire of 21 questions about menopause. Every question can be scored from no complaints to very severe.
Influence of hot flashes on daily life | 6-8 weeks after randomisation and 12 weeks after randomisation
  Influence of hot flashes on daily life will be asked by using a questionnaire: Hot-Flash Related daily interference scale. This 10-item scale measures a woman's perceptions of the degree to which hot flashes interfere with nine daily life activities; the tenth item measures interference with overall quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium